CLINICAL TRIAL: NCT06044012
Title: Double Layer of Buccal Myomucosal Flap and Buccal Pad of Fat for the Closure of Large Oro-antral Fistula
Brief Title: Buccal Myomucosal Flap and Buccal Pad of Fat for the Closure of Oro-antral Fistula
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Ahmed Abdellatif Abdelfatah, Lecturer of oral and maxillofacial surgery, Tanta University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: #R-OS-1-23-3
Record Dates: First submitted 2023-05-08; First posted 2023-09-21 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2024-08

CONDITIONS: Oro-Antral Communication
Keywords: Oro-Antral Fistula; Buccal pad of fat; Myomucosal Flap
MeSH Terms: conditions — Oroantral Fistula

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with large Oro-antral Fistula (Experimental): closure of oro-antral fistula by myomucosal flap and buccal pad of fat
  Interventions: Procedure: Double layer of buccal myomucosal Flap and buccal pad of fat

INTERVENTIONS:
Procedure: Double layer of buccal myomucosal Flap and buccal pad of fat — The buccal myomucosal flap will be harvested from cheek below stenson papilla and will be sutured over buccal pad of fat which will be sutured at palatal mucosa after complete curettage of infected fistulous tract.

SUMMARY:
Oroantral fistula (OAF) is a pathological communication between the oral cavity and the maxillary sinus. A variety of surgical techniques have been developed, with recurrence rates of up to 33%7, mainly due to wound contraction and postoperative infection. To increase the success rates of OAF closure procedures, the use of double-layered closure techniques has developed, but most of these techniques alter the original oral anatomy and may result in significant postoperative morbidity.

ELIGIBILITY:
Inclusion Criteria:

* Large Oro-antral Fistula
* Recent or previously failed closure of oro-antral Fistula

Exclusion Criteria:

* Immuno-supressed patients
* fistulae smaller than 5 mm in size

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-01-01 (Actual)

PRIMARY OUTCOMES:
Healing | 6 months
  The size of fistula will be clinically measured by digital caliper in centimeter for preoperative and postoperative for uneventful wound healing and disappearance of fistula .

SECONDARY OUTCOMES:
infection | 6 months
  fluid level will be measured in cubic centimeter in computed tomography

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Tanta University, Tanta, Egypt